CLINICAL TRIAL: NCT03126734
Title: Effects on Acceptance, Commitment and Awareness of Influence of Parents of Babies With Down Syndrome, After Participation in a Course of Infant Massage. Study on the Spanish Population.
Brief Title: Effects of Infant Massage on Acceptance, Commitment and Conscience of Influence of Parents With Down Syndrome Babies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Elena Piñero Pinto, PhD, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPinto - USeville
Record Dates: First submitted 2017-04-20; First posted 2017-04-24 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Parent-Child Relations
Keywords: Down Syndrome; Acceptance; Commitment; Concience of influence
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The parents of this group will receive 5 sessions of infant massage course (1 per week) between two measurements of the variables
  Interventions: Other: Infant Massage course
- Control Group (No Intervention): The parents of this group will not receive infant massage course (1 per week) between two measurements of the variables. They will receive it after two measurements.

INTERVENTIONS:
Other: Infant Massage course — Infant massage courses consist of 5 sessions. Investigators explain parents how to make an infant massage technique to their babies and which should be the general conditions of the environment.
  This massage is based on the methodology of the International Association of infant massage (IAIM) created by Vimala Schnneider. The courses will make individually.
  Arms: Experimental Group

SUMMARY:
This study aims to analyze whether the course of infant massage serves as a tool to improve acceptance, commitment and awareness of influence of parents of babies with Down syndrome. These variables will be measure before and after the course of infant massage in the experimental group, investigators will make measurements with the same rate in the control group, but they will receive the course after the measurements.

DETAILED DESCRIPTION:
In the present study, investigators propose to study the effects of infant massage in the levels of acceptance, commitment and awareness of influence of parents of babies with Down syndrome. The measuring instrument of acceptance, commitment and awareness of parental influence will be the "This is my baby Interview". Two groups of intervention will be analysed, the experimental, in which parents have participated and applied the knowledge learned in the course of infant massage, and control, which does not receive the infant massage course during the study. Parents and babies of both groups have been evaluated twice, at the beginning of the intervention (pretest) and at the end after five weeks (postest). The study population consists of father or mother of 32 infants with Down syndrome between 4 and 8 months old.

ELIGIBILITY:
Inclusion Criteria:

* Parents with babies with Down Syndrome between 4 and 8 months old.

Exclusion Criteria:

* Parents with babies without Down Syndrome.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
Change from Acceptance | At the start and the end of the study (5 weeks)
  Measure by "This is my baby" Interview

SECONDARY OUTCOMES:
Change fron Commitment | At the start and the end of the study (5 weeks)
  Measure by "This is my baby" Interview

OTHER OUTCOMES:
Change from Conscience of Influence | At the start and the end of the study (5 weeks)
  Measure by "This is my baby" Interview

CONTACTS AND LOCATIONS:
Overall Officials: PIÑERO PINTO, PhD, Principal Investigator — University of Seville
Locations (1):
- Elena Piñero Pinto, Seville, Spain

IPD SHARING:
Plan to Share IPD: No